CLINICAL TRIAL: NCT05029596
Title: Comparative Effectiveness of Heparin Versus Normal Saline in Maintaining Patency of Peripherally Inserted Central Catheter Lines in Oncology Inpatients
Brief Title: Heparin Versus Normal Saline in Peripherally Inserted Central Catheter Lines
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Meredith Allen, Registered Nurse, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STU-2018-0340
Record Dates: First submitted 2021-08-23; First posted 2021-08-31 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Cancer
Keywords: Peripherally Inserted Central Lines; Heparin Flush
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Heparin Group (Active Comparator): Participants will receive the UTSW standard of of care for PICC line maintenance.
  All lumens of PICC line will be flushed w/ Heparin Flush every 8 hours. PICC line will be flushed with 10cc Normal Saline followed by 3cc Heparin Flush after administration of medication, blood products, or blood draws.
  Interventions: Drug: Heparin Group
- Normal Saline Group (Experimental): Participants will receive only Normal Saline for PICC line maintenance. All lumens of PICC line will be flushed every 24 hours with 10cc Normal Saline. PICC line will be flushed with 10cc Normal Saline after administration of medication, blood products, or blood draws.
  Interventions: Drug: Normal Saline Group

INTERVENTIONS:
Drug: Normal Saline Group — A 10cc NS flush will be administered intravenously through the peripherally inserted central line catheter after administration of medication, blood products, and blood draws. In addition the peripherally inserted central line catheter will be flushed intravenously with 10cc Normal Saline every 24 hours.
  Other Names: NS Flush, Normal Saline Flush, 0.9% Normal Saline Flush
  Arms: Normal Saline Group
Drug: Heparin Group — All lumens of PICC line will be flushed w/ Heparin Flush every 8 hours. PICC line will be flushed with 10cc Normal Saline followed by 3cc Heparin Flush after administration of medication, blood products, or blood draws.
  Other Names: Heparin Flush
  Arms: Heparin Group

SUMMARY:
The study team will be performing a study comparing the use of Heparin Flushes vs. Normal Saline Flushes in making sure central lines stay open. The participants will be placed in a group to receive the University of Texas Southwestern Medical Center (UTSW) Standard of Care (control group) for maintaining central lines, or a group to receive Normal Saline Flushes only (experimental group) to keep their central line open. The participants electronic medical record will be reviewed by study team members for the inclusion/exclusion criteria, the participants central line will be assessed by an 11 Blue BMT nurse every 12 hours, and they may be asked questions regarding their medical history during their stay on 11 Blue BMT. If a participant is discharged or transferred off of the 11 Blue BMT unit, they will no longer be included in the study and their central line maintenance will return to the UTSW Standard of Care. Participants in this study may be at risk for central line occlusion (a blood clot) which could require intervention to regain the free flow of fluids and use of the central line. The study team predicts there will be no increase in the rate of line occlusion when using Normal Saline Flushes only to maintain the free flow of fluids through participants central line. The study team also hopes the results of this study will help to improve patient outcomes by decreasing risk of infection, heparin associated complications, and costs.

ELIGIBILITY:
Inclusion Criteria:

* Oncology patients
* Admitted to 11Blue Bone Marrow Transplant Unit at Clements University Hospital University of Texas Southwestern Medical Center
* Ages 18-80 years
* Pre-existing or newly placed PICC line
* PICC line with good blood return (defined as: "brisk blood return of 3cc")
* Flushes without difficulty

Exclusion Criteria:

* Patient less than 18 years of age or greater than 80 years of age
* Refused or unable to give consent to the study
* Patient admitted to the 11Blue BMT unit with any line other than a PICC line, or multiple lines
* Patient admitted to 11Blue BMT for active transplant
* Patient with a coagulopathy diagnosis
* Patient on therapeutic dose of anticoagulants for documented Deep Vein Thrombosis or Pulmonary Embolism
* Patient on inpatient hospice/comfort care
* Patient transferred off 11B BMT unit onto another floor

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Patency | Up to Day 7 of enrollment
  To determine whether or not flushing central lines with normal saline only will maintain free flow through these central lines.

SECONDARY OUTCOMES:
Infection Rate | From Day 1 and up to Day 7 of enrollment
  To determine whether or not removing Heparin Flushes from PICC line maintenance decreases the risk for central line associated infections

CONTACTS AND LOCATIONS:
Overall Officials: Meredith C Allen, BSN, Principal Investigator — University of Texas Southwestern Medical Center; Teresa Phan, Study Chair — University of Texas Southwestern Medical Center; Linda Denke, Study Director — University of Texas Southwestern Medical Center; Kavitha Nair, Study Chair — University of Texas Southwestern Medical Center; Miriam Gonzales, Study Chair — University of Texas Southwestern Medical Center; Ramona Warkola, Study Chair — University of Texas Southwestern Medical Center; Jancy Wilson, Study Chair — University of Texas Southwestern Medical Center
Locations (1):
- Clements University Hospital, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No